CLINICAL TRIAL: NCT03116282
Title: E-alcohol Therapy - an Evaluation of Alcohol Therapy Delivered Via Video Conference
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: TRYG Foundation (Other); Novavi Outpatient Clinics (Unknown)
Responsible Party: Principal Investigator, Kia Kejlskov Egan, PhD student, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 63110-2179
Record Dates: First submitted 2017-03-29; First posted 2017-04-17 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Problematic Alcohol Use
Keywords: e-alcohol therapy; online alcohol treatment; internet-based alcohol treatment; alcohol intervention; video therapy; proactivity
MeSH Terms: interventions — Ethanol; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Conversational therapy via video conference where participants are contacted by an alcohol therapist for the purpose of initiating a course of therapy where participants are not required to show up at a clinic.
  Interventions: Behavioral: E-alcohol therapy
- Control (No Intervention): Treatment as usual where participants receive contact information on their local alcohol treatment facility for the purpose of contacting the facility to initiate a face-to-face course of treatment at the clinic.

INTERVENTIONS:
Behavioral: E-alcohol therapy — Conversational therapy sessions provided via video conference by a professional alcohol therapist.
  Other Names: Electronic alcohol therapy
  Arms: Intervention

SUMMARY:
The study evaluates whether the introduction of e-alcohol therapy (alcohol therapy delivered via video conference) can break with some of the barriers related to alcohol treatment and thereby appeal to people with a problematic alcohol use (Alcohol Use Disorder Test score ≥ 8). The study aims to evaluate the effect of e-alcohol therapy on initiation, treatment compliance and alcohol intake as compared to treatment as usual .

DETAILED DESCRIPTION:
Background: Only a small proportion of those who have a problematic alcohol use receive treatment and compliance is low among the few that undergo treatment. If treatment more easily can be combined with everyday life and break with some of the barriers related to stigma by having a broader appeal, more people with a problematic alcohol use may seek and complete treatment. Alcohol therapy conducted via video conference may be an attractive treatment option and effective in reducing alcohol intake among people with a problematic alcohol use who do not seek traditional treatment.

Objective: The aim of this trial is to evaluate whether people with a problematic alcohol use (Alcohol Use Disorder Test score ≥ 8), who enroll in alcohol therapy delivered via video conference to a greater extent initiate as well as comply with treatment and reduce their alcohol intake compared to people allocated to standard alcohol treatment.

Design: Randomized controlled trial

Participants: 375 Danish citizens above 18 years with a problematic alcohol use (Alcohol Use Disorder Test (AUDIT) score >8).

Intervention: Participants are randomized to one of two groups:

1. Conversational therapy via video conference where participants are contacted by an alcohol therapist for the purpose of initiating a course of treatment where participants are not required to show up at a clinic.
2. Treatment as usual where participants receive contact information on their local alcohol treatment facility for the purpose of contacting the facility to initiate a face-to-face course of treatment at the clinic.

The allocation of participants to the intervention will be 1:1 to the intervention and the control group.

Methods: Data will be collected by questionnaire at baseline, 3 months and 12 months post randomization. Analyses will be intention to treat. Subgroup analysis will be conducted in relation to personal and demographic characteristics.

Process evaluation will be performed using a combination of questionnaires and qualitative interviews with participants, therapists and management at the clinics.

ELIGIBILITY:
Inclusion Criteria:

- Problematic alcohol consumption (Alcohol Use Disorder Test score ≥ 8)

Exclusion Criteria:

* Not legally able and willing to provide informed consent
* No provision of a functional e-mail address
* No provision of municipality of residence and phone number
* No access to a personal computer equipped with functional camera, audio equipment, and Internet access.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Initiation of treatment (completion of one session) | 3 months post randomization
  25% higher completion of one treatment session
Initiation of treatment (completion of one session) | 12 months post randomization
  25% higher completion of at least one treatment sessions
Compliance (completion of at least 3 sessions) | 3 months post randomization
  25% higher completion of at least three treatment sessions
Compliance (completion of at least 3 sessions) | 12 months post randomization
  25% higher completion of at least three treatment sessions
Total weekly alcohol intake (measured by Timeline follow back) | 3 months post randomization
  Higher reduction in total weekly alcohol intake (measured by Timeline follow back) (5 units)
Total weekly alcohol intake (measured by Timeline follow back) | 12 months post randomization
  Higher reduction in total weekly alcohol intake (measured by Timeline follow back) (5 units)

SECONDARY OUTCOMES:
Weekly alcohol intake below national guidelines | 3 and 12 months post randomization
  20% increase in participants reporting a weekly alcohol intake below the national high risk drinking limits.
Weekly number of heavy drinking days | 3 and 12 months post randomization
  Lower number of weekly heavy drinking days (5+ units in one occasion)
Weekly drinking days | 3 and 12 months post randomization
  Lower number of weekly drinking days
Problematic drinking | 12 months post randomization
  Lower Alcohol Use Disorder Test score
Quality of life | 3 and 12 months post randomization
  Higher quality of life as measured by the 'Cantril Ladder'

CONTACTS AND LOCATIONS:
Overall Officials: Janne Tolstrup, Professor, Study Director — University of Southern Denmark; Ulrik Becker, Professor, Study Director — University of Southern Denmark
Locations (1):
- National Institute of Public Health, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Egan KK, Becker U, M Ller SP, Pisinger V, Tolstrup JS. Effectiveness of proactive video therapy for problematic alcohol use on treatment initiation, compliance, and alcohol intake: a randomised controlled trial in Denmark. Lancet Digit Health. 2024 Jun;6(6):e418-e427. doi: 10.1016/S2589-7500(24)00067-0. PMID 38789142